CLINICAL TRIAL: NCT07314736
Title: Stakeholders of Rare Diseases Informing Values In Neuroethics
Status: Not yet recruiting | Type: Observational
Sponsor: St. Jude Children's Research Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: STRIVE
Record Dates: First submitted 2025-12-16; First posted 2026-01-02 (Actual); Last update posted 2026-01-02 (Actual); Status verified 2025-12

CONDITIONS: Rare Disorder; Disorder, Neurologic
Keywords: Rare Neurological Disorders (RND); Stakeholders; Patient Participant; Caregiver; Other Family; Non-Family Stakeholder
MeSH Terms: conditions — Rare Diseases; Nervous System Diseases

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Primary Caregivers/Patients: Primary caregivers of children/young adults (age 21 or younger) and patients (age 25 or younger) diagnosed with a super-rare, catastrophic neurologic disorder without definitive FDA-approved treatment.
- Other Family Stakeholders: Siblings (13 years or older) and extended family members (e.g., grandparents) and primary caregivers who prefer not to participate in the longitudinal component
- Non-Family Stakeholders: Non-family stakeholders involved in the clinical care or investigational treatments of children with catastrophic illnesses.

SUMMARY:
The purpose of this research study is to learn more about the perspectives of key stakeholders-patients, families, healthcare providers, and researchers-on the ethical challenges of small-scale, personalized treatment trials for rare neurological diseases (RND).

DETAILED DESCRIPTION:
Primary Objectives

* To utilize semi-structured interviews to identify key stakeholder preferences and gather recommendations for the ethical conduct of n-of-few approaches in pediatric patients with rare neurological diseases (RND).
* Identify key challenges and best practices for informed consent and communication strategies for personalized interventions in pediatric RND trials.
* To develop a best practice framework for the ethical conduct of research involving personalized interventions for children with catastrophic RND.

Secondary Objectives

* To use surveys to quantitatively measure trust in health care providers and medical researchers, quality of life, and resilience in families of a patient or patients with an RND.
* To elicit feedback from patients and families on their perceived utility of existing patient reported outcome (PROs) measures relevant to capturing their illness experience and needs.

This study will employ a mixed-methods approach to comprehensively understand the perspectives of families and non-family stakeholders regarding personalized research programs in super-rare, catastrophic neurologic disorders. The study will utilize validated surveys, semi-structured interviews, and focus groups.

Group 1: Primary Caregivers/Patients (Longitudinal Approach)

* Participants will complete validated quality-of-life inventories at baseline and once-to-twice per year over the study period.
* Semi-structured interviews will be conducted at the time of enrollment, then approximately every 6 months through the end of the study period, focusing on:

  * Views on a priori-defined research ethics topics.
  * Understanding the family's illness experience and any significant changes since the previous interview.
  * Reflective recaps of previous interviews to identify shifts in attitudes.

Group 2: Other Family Stakeholders (Cross-Sectional Approach)

* This group will participate in single interviews or focus groups, as determined by participant choice. Participants will be referred to study team by Group 1 participants and will be interviewed after their relative in Group 1 has completed at least one interview. They will provide insights into how families apply the concepts of the Belmont Report (e.g., autonomy and justice) to their experiences and define "benefit" and "risk" in the context of personalized treatments.
* This portion of the study will focus on patient-reported outcomes (PROs) that are meaningful to families.

Group 3: Non-Family Stakeholders

* Semi-structured interviews, focus groups, and listening sessions will be conducted to explore ethical best practices and potential pitfalls in delivering n-of-few therapies.

ELIGIBILITY:
Inclusion Criteria:

Group 1 (Parental Caregiver and Patient Participants)

* Parental/primary caregiver with a child who has a genetic diagnosis of an ultrarare disorder with pediatric onset, or a clinical diagnosis with a suspected genetic etiology.
* Child is under 21 years of age at the time of enrollment.
* Child has an expected survival of at least one year following study enrollment.
* Patients (age ≤ 25 years) with a genetic diagnosis of an ultrarare disorder with pediatric onset, or clinical diagnosis with suspected genetic etiology.
* Willingness to provide verbal informed consent (or assent, as appropriate) to participate

Group 2 (Other Family)

* Family member of a Group 1 participant who plays an active role in the child's life or care.
* Includes siblings (≥ 13 years of age), grandparents, or other non-primary caregivers directly affected by the child's diagnosis.
* Demonstrated familiarity with the child's medical and family experience.
* Willingness to provide verbal informed consent (or assent, as appropriate) to participate.

Group 3 (Non-Family Stakeholders)

* Individuals currently engaged, or recently active, in clinical care, research, advocacy or policy work related to pediatric-onset rare genetic disorders.
* May include clinicians (e.g., neurologists, genetic counselors, nurses, child-life specialists, home-health staff), members of patient-advocacy organizations, institutional-review-board (IRB) members, payers, sponsors, funders, or representatives of hospital systems or regulatory agencies.
* Willingness to provide verbal informed consent to participate in semi-structured interviews or focus groups

Exclusion Criteria:

* Limited English proficiency
* Unable to complete the survey materials or complete the interviews in English.
* Inability or unwillingness of research participant to give verbal informed consent (in English)
* • Condition or chronic illness, which in the opinion of the PI/Co-I, makes participation unsafe or untenable (i.e., cognitive impairment, concurrent acute morbidity).

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Those who meet the Eligibility Criteria and agree to participate.
Sampling Method: Non-Probability Sample
Enrollment: 385 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2031-01 (Estimated); Study Completion 2031-01 (Estimated)

PRIMARY OUTCOMES:
Identifying key stakeholder preferences and recommendations for the ethical conduct of n-of-few approaches in pediatric patients with rare neurological diseases (RND) utilizing semi-structured interviews | At baseline and every 6 months until end of study, approximately 5 years (Group 1); Once, within 60 days of enrollment (single interview per Group 2 and 3 participant)
  Semi-structured interviews will be analyzed using MAXQDA software to identify themes though a systematic and standardized process. A deductive approach willl be used to formulate initial codes based on research questions and interview guides developed. Additional themes and codes will be developed using an inductive approach where new codes are allowed to emerge after review of the transcripts by three study team members trained in content analysis. To compensate for the multiple appearance of a code in a single interview, the percentage of patients for whom the code appeared will be tallied. Codes will be grouped and identified as a theme that captures the shared meaning. The definitions of each of the combined codes will be compared to arrive at a final definition for each theme. As with the codes, the frequency of occurrence of each theme and the percentage of patients to which each theme applied will be tallied, as well as inter-rater reliability.
Identify key challenges and ethics-informed best practices for the development and implementation of personalized or n-of-few genomic interventions for rare and catastrophic pediatric disorders. | At baseline and every 6 months until end of study, approximately 5 years (Group 1); Once, within 60 days of enrollment (single interview per Group 2 and 3 participant)
  Semi-structured interviews will be analyzed using MAXQDA software to identify themes though a systematic and standardized process. A deductive approach will be used to formulate initial codes based on research questions and interview guides developed. Additional themes and codes will be developed using an inductive approach where new codes are allowed to emerge after review of the transcripts by three study team members trained in content analysis. To compensate for the multiple appearance of a code in a single interview, the percentage of patients for whom the code appeared will be tallied. Codes will be grouped and identified as a theme that captures the shared meaning. The definitions of each of the combined codes will be compared to arrive at a final definition for each theme. As with the codes, the frequency of occurrence of each theme and the percentage of patients to which each theme applied will be tallied, as well as inter-rater reliability.
To develop a best practice framework for the ethical conduct of research involving personalized interventions for children with catastrophic genetic disorders of childhood onset. | The panel will meet quarterly, beginning formal framework development in Year 3 until study completion, approximately 5 years.
  An interdisciplinary advisory panel of approximately 20 expert partners will be established. The panel will be presented with clearly defined problems-on elements of respect for persons (informed consent, parental autonomy), beneficence (risk-benefit assessments), justice (fair subject selection, equity) and research obligations, among others-which will be reframed to them from multiple perspectives (from results of Objective 1 and 2). The working group will engage in decisional analysis, identifying and evaluating value trade-offs through moral discussion and consensus. This iterative process of integrating normative content with empirical findings will then lead to practical recommendations, optimizing positives and minimizing negatives.

SECONDARY OUTCOMES:
To elicit feedback from patients and families on their perceived utility of existing patient reported outcome (PROs) measures relevant to capturing their illness experience and needs. | At baseline and every 6 months until end of study, approximately 5 years
  Parent and Patient-Reported Outcomes (PROs) will be quatified using the Patient Specific Functional Scale (PSFS). The parents or patient will identify five important activities that their child is having difficulty with as a result of their condition. The parent rates difficulty on an 11-point numerical scale (0= unable to perform the activity: 10= able to perform activity. The average score for the five activities is the PSFS score. (ages one month-21 years) Higher scores indicate better functional ability in patient-identified, meaningful daily activities; lower scores indicate greater functional limitation in those activities. Since the PSFS is individualized, not norm-referenced, scores are meant to track change within the same child over time, rather than functioning as a tool for interpersonal comparison.
Human Connection Scale | Baseline, then approximately annually during the study period, approximately 5 years
  Caregiver trust in the child's health care provider will be assessed using the Human Connection Scale. This instrument evaluates how caregivers experience meaningful relationships within the health care context, including perceived empathy, understanding, emotional support, and attentiveness of the provider. Items are rated on a Likert-type scale reflecting agreement, confidence, or frequency and are summed to produce a total human connection score. Higher scores indicate greater perceived trust and stronger caregiver-provider relationships. Trust is examined as a factor that may influence caregiver willingness to pursue highly investigational treatments.
Trust in Medical Researchers Scale | Baseline, then approximately annually during the study period, approximately 5 years.
  Caregiver trust in medical researchers and the research process will be measured using the Trust in Medical Researchers scale. This instrument assesses perceptions of researcher honesty, competence, transparency, and respect for participants, reflecting caregivers' experiences of meaningful relationships within the research context. Items are rated on a Likert-type scale and summed to generate an overall trust score. Higher scores indicate greater trust in medical researchers and the research enterprise.
Caregiver Resilience (Connor-Davidson Resilience Scale) | Baseline, then approximately every 6 months during the study period, approximately 5 years
  Caregiver resilience in the context of a child's catastrophic illness will be measured using the Connor-Davidson Resilience Scale (CD-RISC). The CD-RISC consists of 25 items assessing domains including persistence, adaptability, sense of control, optimism, coping with stress, burden, uncertainty, and fears. Items are rated on a 5-point Likert scale from 0 to 4 and summed to produce a total resilience score. Higher scores represent greater caregiver resilience.
Baseline, then approximately every 6 months during the study period | Baseline, then approximately every 6 months during the study period, approximately 5 years.
  Caregiver support needs will be assessed using the Caregiver Support Assessment Tool (CSNAT). The CSNAT is a 14-item instrument designed to identify caregiver needs across two domains: support required to enable caregiving activities and support required for the caregiver's own well-being. Each item is rated on a 4-point scale ranging from "no more support needed" to "very much more support needed." Responses are used to generate a profile of unmet support needs across domains, with higher ratings indicating greater unmet need.
Infant Health-Related Quality of Life (PedsQL Infant Module) | Baseline, then approximately every 6 months during the study period, approximately 5 years
  Infant health-related quality of life will be measured using the PedsQL Infant Module. This parent-proxy instrument includes 36 items for infants aged 1-12 months and 45 items for infants aged 13-24 months. Subscales assess physical functioning, physical symptoms, emotional functioning, social functioning, and cognitive functioning. Items are rated on a Likert scale, reverse scored, and linearly transformed to a 0-100 scale. Domain and total scores are calculated as averages of item scores, with higher scores indicating better quality of life.
Child and Adolescent Health-Related Quality of Life (PedsQL v4.0 Generic Core Scales) | Baseline, then approximately every 6 months during the study period, approximately 5 years
  Health-related quality of life in children and adolescents will be assessed using the PedsQL v4.0 Generic Core Scales. This 23-item instrument includes subscales measuring physical, emotional, social, and school functioning. Items are rated on a Likert scale, reverse coded, and transformed to a 0-100 scale. Domain and total scores are calculated as averages of item scores, with higher scores indicating better quality of life. Patient self-report and parent-proxy versions are used based on age. Items not meeting internal consistency thresholds will be reported descriptively.
Neuromuscular Disease-Specific Quality of Life (PedsQL 3.0 Neuromuscular Module) | Baseline, then approximately every 6 months during the study period, approximately 5 years
  Disease-specific quality of life will be measured using the PedsQL 3.0 Neuromuscular Module. This 25-item instrument includes three domains: neuromuscular disease symptoms and impacts, communication about illness, and family resources. Items are rated on a Likert scale, reverse coded, and transformed to a 0-100 scale. Domain and total scores are calculated as averages of item scores, with higher scores indicating better disease-specific quality of life and family functioning. This measure will be completed only by participants with neuromuscular conditions.

CONTACTS AND LOCATIONS:
Overall Officials: Liza M. Johnson, MD, MPH, MSB, Principal Investigator — St. Jude Children's Research Hospital
Locations (1):
- St. Jude Children's Research Hospital, Memphis, Tennessee, United States

REFERENCES:
- See also: St. Jude Children's Research Hospital — http://www.stjude.org
- See also: Clinical Trials Open at St. Jude — http://www.stjude.org/protocols